CLINICAL TRIAL: NCT03631108
Title: Feasibility Study and Preliminary Application Study on Noninvasive Iris Optical Coherence Tomography Angiography (OCTA)
Brief Title: Feasibility Study and Preliminary Application Study on Iris OCTA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018KY181
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Conjunctivitis; Glaucoma; Myopia; Diabetic Retinopathy; Retinal Detachment; Retinal Neovascularization, Unspecified; Uveitis
Keywords: Iris Vessel; OCTA
MeSH Terms: conditions — Conjunctivitis; Glaucoma; Myopia; Diabetic Retinopathy; Retinal Detachment; Retinal Neovascularization; Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal Population: Normal population with different gender, different age different, different blood pressure, different ocular pressure, etc.
  All participants will underwent imaging using the OCTA system (Zeiss) with the anterior segment optical adaptor lens.
- Patients with common ophthalmic diseases: (1) conjunctivitis; (2) glaucoma; (3) childhood myopia; (4) uveitis; (5) diabetic retinopathy; (6) retinal detachment; (7) fundus neovascularization.
  All patients will underwent imaging using the OCTA system (Zeiss) with the anterior segment optical adaptor lens.
- Patients using eye drops: (1) conjunctivitis patients treated with levofloxacin antibiotics; (2) glaucoma patients treated with prostaglandins, adrenaline or receptor blockers drugs; (3) childhood myopia patients treated with atropine drugs; (4) uveitis patients treated with hormones treatment. (5) diabetic retinopathy patients treated with vasodilator.
  All patients will underwent imaging using the OCTA system (Zeiss) with the anterior segment optical adaptor lens before and after eyedrops.
  Interventions: Diagnostic Test: OCTA (ZEISS)
- Ocular surgery patients: (1) cataract, phacoemulsification + intraocular lens implantation; (2) glaucoma, iridectomy; (3) fundus neovascularization, intraocular injection of anti-VEGF; (4) diabetic retinopathy, vitrectomy.
  All patients will underwent imaging using the OCTA system (Zeiss) with the anterior segment optical adaptor lens before and after surgery.
  Interventions: Diagnostic Test: OCTA (ZEISS)

INTERVENTIONS:
Diagnostic Test: OCTA (ZEISS) — All participants will underwent imaging using the OCTA system (Zeiss) with the anterior segment optical adaptor lens.
  Groups: Ocular surgery patients; Patients using eye drops

SUMMARY:
All participants will underwent imaging using the OCTA system (Zeiss) with the anterior segment optical adaptor lens. The main outcomes are iris blood flow density and vascular density.

DETAILED DESCRIPTION:
1. Feasibility study of iris OCTA technology
2. Establishment of iris OCTA database in normal population and analysis of related factors: (1) different sex; (2) different age; (3) different myopic diopter; (4) 24-hour diurnal changes from morning to night; (5) before and after mydriasis; (6) different blood pressure; (7) different intraocular pressure; (8) different blood glucose; (9) before and after exercise. (10) drinking water, tea, coffee and red wine.
3. Analysis of iris OCTA data related to eye diseases:(1) conjunctivitis; (2) glaucoma; (3) childhood myopia; (4) uveitis; (5) diabetic retinopathy; (6) retinal detachment; (7) fundus neovascularization.
4. Influence of commonly used ophthalmic drops on iris OCTA data. Observe the difference of iris OCTA test data before and after treatment: (1) conjunctivitis treated with levofloxacin antibiotics; (2) glaucoma treated with prostaglandins, adrenalines and receptor blockers; (3) childhood myopia treated with atropine drugs (4) uveitis treated with hormonal drugs. (5) diabetic retinopathy treated with vasodilator.
5. Effect on iris OCTA data before and after ophthalmic surgery. (1) cataract, phacoemulsification + intraocular lens implantation; (2) glaucoma, iridectomy; (3) fundus neovascularization, intraocular injection of anti-VEGF; (4) diabetic retinopathy, vitreous surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and ophthalmological patients who can understand and agree to cooperate this study will be included.

Exclusion Criteria:

* Patients who can not cooperate with the examination.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Shanghai and patients from Shanghai Eye Hospital will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Iris Vessel Geometric Characteristics | 0:00 8:00 14:00 20:00
  Iris vascular density and neovascular density

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cui L, Xiao Y, Xiang Z, Chen Z, Yang C, Zou H. Study on the correlation between iris blood flow, iris thickness and pupil diameter in the resting state and after pharmacological mydriasis in patients with diabetes mellitus. BMC Ophthalmol. 2024 Feb 2;24(1):52. doi: 10.1186/s12886-024-03322-y. PMID 38308203
- [Derived] Jia Y, Xue W, Tong X, Wang Y, Cui L, Zou H. Quantitative analysis and clinical application of iris circulation in ischemic retinal disease. BMC Ophthalmol. 2021 Nov 15;21(1):393. doi: 10.1186/s12886-021-02165-1. PMID 34781913